CLINICAL TRIAL: NCT03826589
Title: Avelumab With Axitinib in Persistent or Recurrent Cervical Cancer After Platinum-based Chemotherapy - a Proof-of-concept Study (ALARICE Study)
Brief Title: Avelumab With Axitinib in Persistent or Recurrent Cervical Cancer After Platinum-based Chemotherapy
Acronym: ALARICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ka-Yu Tse, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI224183 / UW 18-417
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Avelumab; Axitinib
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — avelumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avelumab and Axitinib (Experimental): * Avelumab: IV treatment; administered at 10 mg/kg IV every two weeks in a 4-weekly cycle up to 12 cycles or until disease progression or intolerable side effects (whichever occurs first)
  * Axitinib: Oral treatment; administered at 5 mg PO BID in a 4-weekly cycle up to 12 cycles or until disease progression or intolerable side effects (whichever occurs first)
  Interventions: Drug: Avelumab; Drug: Axitinib

INTERVENTIONS:
Drug: Avelumab — an anti-programmed cell death ligand 1
  Other Names: Bavencio
Drug: Axitinib — a tyrosine kinase inhibitor that also inhibits VEGF receptor 1-3, c-KIT and PDGFR
  Other Names: Inlyta

SUMMARY:
This is a single-arm, Simon's 2-stage, proof-of-concept trial. The aim is to evaluate the efficacy and safety of avelumab with axitinib in patients with persistent or recurrent cervical cancer following platinum-based chemotherapy. The study hypothesis is that the combination of avelumab and axitinib can significantly improve the objective response rate (ORR) with acceptable toxicity compared to traditional chemotherapy.

DETAILED DESCRIPTION:
Cervical cancer is the fourth commonest female cancer in the world. When there is distant metastasis or recurrence, platinum-based chemotherapy is the usual treatment option. Once this first-line chemotherapy fails, the prognosis is dismal. Various second-line agents including second-line chemotherapy agents and immune checkpoint inhibitors have unsatisfactory response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years old.
2. Patients must have histologically confirmed cervical cancer, either squamous cell, adenocarcinoma or adenosquamous, that is either persistent or recurrent after at least one prior course of platinum-based chemotherapy. The platinum used in concurrent chemo-irradiation is not counted.
3. Patients should not be amenable to further surgery or radiotherapy except for the purpose of symptomatic relief.
4. Patients should have ECOG performance score 0 to 2.
5. Patients must have at least one target lesion by the RECIST 1.1 criteria.
6. Prior chemotherapy must have been completed at least 3 weeks before study drug administration, and all AEs have either returned to baseline or stabilized.
7. Prior systemic radiation therapy must have been completed at least 4 weeks before study drug administration. Prior focal radiotherapy must have completed at least 2 weeks before study drug administration.
8. Patients must have recovered from any major surgery that has been done at least 4 weeks before study drug administration.
9. Patients must have adequate bone marrow, renal, hepatic, thyroid and neurological function.
10. Patients should be willing to have blood tests where the blood will be used for biomarker studies.
11. Formalin-fixed, paraffin-embedded (FFPE) archival tumor specimens of the primary tumors, should be available during screening. Alternatively, 15 unstained slides (6 minimum) will be acceptable.
12. Patients should agree for de novo biopsy if the tumors are at the cervix or vagina, or any other sites that are easy and safe to be biopsied. Tumors will be used for biomarker studies.
13. Patients who have childbearing potential should practice highly effective contraception throughout the study until at least 30 days after completion of the treatment

Exclusion Criteria:

1. Patients with concurrent malignancy within five years (except for basal or squamous cell skin cancer or in-situ breast cancer) are excluded.
2. Patients who have history of autoimmune diseases or other diseases requiring systemic steroid are excluded.

   Patients with vitiligo, type I diabetes mellitus, resolved asthma or atopy, stable autoimmune thyroid disease, eczema, psoriasis not requiring systemic treatment*, or not expected to recur in the absence of an external trigger are permitted to enroll.
3. Patients with the following past significant medical history in the last six months are excluded, such as pneumonitis, active or chronic viral hepatitis, cirrhosis, and inherited liver disease, myocardial infarction, unstable angina, unstable cardiac arrhythmia or clinically significant valvular heart diseases, CTCAE Grade 2 or greater peripheral vascular disease, active brain metastases or leptomeningeal metastases, uncontrolled seizures, subarachnoid hemorrhage, thromboembolic events.
4. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days of the start of treatment are excluded. Inhaled, local or topical steroids, systemic corticosteroids at physiologic doses, steroid used as pre-medication are allowed.
5. Patients with severe gastrointestinal conditions such as evidence of bowel obstruction or uncontrolled diarrhea in the last 4 weeks prior to enrollment, or history of inflammatory bowel disease, are not eligible.
6. Patients with uncontrolled hypertension (systolic >160mmHg or diastolic > 110mmHg) despite medication, active bleeding, bone fracture, unhealed wounds, clinically significant proteinuria (> 2g of protein over 24 hours), are excluded.
7. Patients with unhealed wounds include abdominal or pelvic fistula, gastrointestinal perforation or intra-abdominal abscess are excluded.
8. Patients having had severe infections within 4 weeks prior to the start of treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, and those who have active infection requiring systematic treatment, are excluded.
9. Patents with active tuberculosis, history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) are excluded.
10. Patients who have suicidal ideations or behaviors requiring psychiatric intervention within 3 months prior to the start of treatment are excluded.
11. Patients who have history of severe (CTCAE Grade 3 or above) hypersensitivity reaction to any investigational products or any component in its formulations, and any monoclonal antibody, are excluded.
12. Patients who have known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the avelumab formulation.
13. Patients who have persisting toxicities related to previous therapy (NCI CTCAE v 5.0 Grade >1) are excluded. However, alopecia, Grade 2 or less sensory neuropathy, or other toxicities of Grade 2 or below that do not constitute a safety risk according to the investigators' judgment, are allowed.
14. Patients who have received prior immunotherapy, such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, are excluded.
15. Patients who have received axitinib before are excluded.
16. Patients who received other anti-angiogenics within the last 6 months are excluded.
17. Patients with prior allogeneic stem cell or solid organ transplantation are excluded.
18. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or at least 5 half-lives (whichever is longer) before the start of treatment, or during the course of this trial, is not allowed.
19. Use of any live attenuated vaccines against infectious diseases (e.g. influenza, varicella, etc.) within 4 weeks (28 days) of the start of treatment and during the study therapy is not allowed.
20. Patients with major operation within 28 days or open biopsy within 7 days before enrolment are not eligible.
21. Patients planned to have major surgery during the course of the study are excluded.
22. Patients who are pregnant or breastfeeding are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of patients who have a CR or PR to the study drugs.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  The time from first dose of trial medication to first documentation of objective tumor progression (PD) or to death due to any cause, whichever occurs first.
Overall survival | Up to 2 years
  Overall survival is defined as the time from first dose of trial medication to date of death due to any cause.
Objective tumor response rate | Up to 2 years
  Objective tumor response rate according to the immune-related ResponseCriteria Derived from RECIST 1.1 (irRECIST)
Disease control rate at 12 weeks | Up to 2 years
  Disease control rate at 12 weeks including complete response (CR), partial response (PR), stable disease (SD)
Duration of response | Up to 2 years
  Duration of response and duration of clinical benefit including CR, PR and SD
Rates of abnormal laboratory values and/or adverse events that are related to the treatment drugs | Up to 2 years
  Treatment-related adverse events classified by CTCAE version 5.0 and laboratory safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yu Tse, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Undecided